CLINICAL TRIAL: NCT02793011
Title: Does Dexamethasone Reduce Postoperative Pain in Pediatric Tonsillectomy Patients?
Brief Title: Dexamethasone and Post-tonsillectomy Pain in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Olubukola Nafiu, Assistant Professor of Anesthesiology, University of Michigan Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00084860; 5K23GM104354 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-06-08 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Pediatric Post-tonsillectomy Pain
MeSH Terms: interventions — Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Liquid or capsule dexamethasone - to be taken orally the evening before scheduled tonsillectomy with or without adenoidectomy
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo liquid or capsule to be taken orally the evening before scheduled tonsillectomy with or without adenoidectomy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Oral dexamethasone elixir (0.5mg/ml or 4 mg/ml) mixed with Ora-sweet or simple syrup to mask the taste. Or 1 mg or 4 mg dexamethasone capsules if age appropriate
  Other Names: corticosteroid
  Arms: Dexamethasone
Drug: Placebo — Placebo liquid (Ora-sweet or simple syrup) or Placebo capsule
  Arms: Placebo

SUMMARY:
The investigators will use a prospective randomized, controlled design utilizing a single preoperative dose of oral dexamethasone or placebo to achieve these specific aims:

* Specific Aim 1: To evaluate the potential for a single preoperative dose of oral dexamethasone administered the night before surgery to reduce the incidence and severity of early post tonsillectomy pain (PTP) in children
* Specific Aim 2: To prospectively evaluate differences in early PTP experience between overweight/obese children and their lean peers.
* Specific Aim 3: To determine whether circulating inflammatory markers are strongly linked to PTP severity in children and whether they could be potential contributors to the higher pain experienced by overweight/obese children following Tonsillectomy and or Adenoidectomy.

DETAILED DESCRIPTION:
(See brief summary as well)

The study will serve as a vehicle for a three-pronged approach (clinical observation, biological basis and therapeutic intervention) reflects the applicants professional interest in translational pediatric obesity research If the investigators find that BMI-dependent disparity exists in Post Tonsillectomy Pain (PTP) and that preoperative down regulation of inflammatory response with one preoperative dose of corticosteroids reduces PTP, our findings should ultimately lead to improved postoperative pain management of pediatric PTP especially in obese children.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for tonsillectomy and/or adenoidectomy at University of Michigan, C. S. Mott Children's Hospital

Exclusion Criteria:

* Known hypersensitivity to dexamethasone
* Developmental delay
* Taking chronic analgesics
* Taking chronic systemic steroids
* Treatment with steroids in last 30 days
* Cushings or Prader-Willi or Nephrotic Syndromes
* Diabetes Mellitus

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2016-06; Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
Incidence of moderate/severe pain(>/= 4 of 10 using the Wong-Baker faces Scale) during recovery room stay | 0-8 hours postoperatively
  Subjects will be evaluated in the Post Anesthesia Care Unit (PACU) until discharge home or to the unit.

SECONDARY OUTCOMES:
Proportion of patients requiring analgesic intervention in the PACU will differ by BMI category (normal, overweight and obese). | 0-8 hours postoperatively
  Subjects will be evaluated in the Post Anesthesia Care Unit (PACU) until discharge home or to the unit.
Bivariate association between BMI (in Kg/m2) and serum values of inflammatory markers (CRP, TNF-alpha and IL-6) will be computed. | 0-8 hours postoperatively
  Subjects will be evaluated in the Post Anesthesia Care Unit (PACU) until discharge home or to the unit.

CONTACTS AND LOCATIONS:
Overall Officials: Olubukola Nafiu, MD, Principal Investigator — University of Michigan, CS Mott Children's Hospital, Dept of Otolaryngology
Locations (1):
- University of Michigan C.S. Mott Children's Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No